CLINICAL TRIAL: NCT03374202
Title: VRC 603: A Phase I Dose-Escalation Study of the Safety of AAV8-VRC07 (VRC-HIVAAV070-00-GT) Recombinant AAV Vector Expressing VRC07 HIV-1 Neutralizing Antibody in Antiretroviral-Treated, HIV-1 Infected Adults With Controlled Viremia
Brief Title: Safety and Tolerability of AAV8 Delivery of a Broadly Neutralizing Antibody in Adults Living With HIV: a Phase 1, Dose-escalation Trial
Acronym: VRC 603
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 180030; 18-I-0030
Record Dates: First submitted 2017-12-14; First posted 2017-12-15 (Actual); Results first posted 2023-10-25 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: HIV-1 Infected Adults With Controlled Viremia
Keywords: ARV Therapy; Broadly Neutralizing; Gene Transfer; Monoclonal Antibody; AAV8

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: AAV8-VRC07 (5 x 10^10 vg/kg IM) (Experimental): AAV8-VRC07 (5 x 10^10 vg/kg) administered by intramuscular (IM) injection (Day 0)
  Interventions: Genetic: VRC-HIVAAV070-00-GT (AAV8-VRC07)
- Group 2: AAV8-VRC07 (5 x 10^11 vg/kg IM) (Experimental): AAV8-VRC07 (5 x 10^11 vg/kg) administered by IM injection (Day 0)
  Interventions: Genetic: VRC-HIVAAV070-00-GT (AAV8-VRC07)
- Group 3: AAV8-VRC07 (2.5 x 10^12 vg/kg IM) (Experimental): AAV8-VRC07 (2.5 x 10^12 vg/kg) administered by IM injection (Day 0)
  Interventions: Genetic: VRC-HIVAAV070-00-GT (AAV8-VRC07)

INTERVENTIONS:
Genetic: VRC-HIVAAV070-00-GT (AAV8-VRC07) — AAV8-VRC07 is a recombinant AAV vector expressing a HIV-1 CD4 binding site-specific neutralizing antibody, VRC07

SUMMARY:
Background:

The Human Immunodeficiency Virus (HIV) attacks the immune system. Scientists have created a gene that could be transferred to the cells of people with HIV. The gene should tell the cells to make an antibody called VRC07. This antibody fights HIV. The VRC07 gene is packaged into a man-made version of a virus called AAV8.

Objectives:

To see if AAV8-VRC07 is safe. To study if it causes cells to produce the VRC07 antibody.

Eligibility:

Adults ages 18-65 who are HIV infected but in general good health and have been taking the same HIV medicine for at least 3 months

Design:

Participants were screened in a different protocol.

Participants received the study product on day 1. It was injected one or more times in the upper arm or thigh using a needle. Participants weight was measured to calculate the dose.

Women may have had a pregnancy test.

For 7 days after getting the study product, participants checked their temperature with a thermometer. They noted any symptoms in an electronic or paper diary.

Participants will have study visits. At each one, they will have a physical exam and medical history. They will have blood drawn and may have saliva collected.

The study visit schedule is as follows:

For 12 weeks: 1 visit a week

For the next 12 weeks: 1 visit every other week

Then about 1 visit a month

After 1 year in the study: a visit every 6 months for the next 4 years.

Total study participation is 5 years.

DETAILED DESCRIPTION:
Design: This is a Phase I study of the safety and tolerability of AAV8-VRC07 (VRC-HIVAAV070-00-GT) expressing VRC07 human monoclonal antibody with broad HIV-1 neutralizing activity in HIV-1 infected adults. It is a dose-escalation study to examine pharmacokinetics of VRC07 expression following intramuscular (IM) administration of AAV8-VRC07 in participants on anti-retroviral therapy (ARV). The hypotheses are: 1) AAV8-VRC07 will be safe for human administration and will not elicit hypersensitivity or anti-drug antibody (ADA) to VRC07; and 2) intramuscular delivery of AAV8-VRC07 will result in production of biologically active VRC07 antibody at a concentration in serum that is measurable and safe.

Description: AAV8-VRC07 was developed by VRC, NIAID, NIH, and manufactured by the Clinical Vector Core, Center for Cellular and Molecular Therapeutics, The Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania (PA). It is composed of an AAV8 recombinant vector expressing genes encoding the heavy and light chains of the VRC07 monoclonal antibody. AAV8-VRC07 was supplied at 2.84 x 10^13 vector genomes (vg)/mL.

Participants: HIV-1 infected adult volunteers (18 to 65 years old) on a stable antiretroviral regimen for more than or equal to 3 months, with controlled viremia, under the care of a physician, and without additional clinically significant medical conditions.

Study Plan: There are 3 dose escalation groups. Sequentially enrolled participants were assigned to the dosage level being evaluated at the time of enrollment. All injections were administered intramuscularly (IM) by needle and syringe. Cumulative safety data were reviewed weekly by a Protocol Safety Review Team (PSRT) that included an Independent Safety Monitor (ISM) while injections were being administered. Safety, including reactogenicity and unsolicited adverse events (AEs), laboratory findings, pharmacokinetics, and VRC07 antibody levels in blood were assessed after the injection and summarized for an interim analysis at 4 weeks post injection. The second participant in each dose group was injected after the 4 weeks safety assessment for the first participant. Decisions regarding dose escalation and participant enrollments were based on safety data and the VRC07 concentration in blood at 4 weeks after product administration. The pharmacokinetics of VRC07 at each dose level was evaluated to determine the dose that would result in antibody production that achieves at least 50 mcg/mL VRC07 concentration in serum at 4 weeks post injection with a target set point of more than or equal to 5 mcg/mL at 12 weeks post injection.

ELIGIBILITY:
INCLUSION CRITERIA:

A volunteer must have met all of the following criteria:

* Able and willing to complete the informed consent process.
* 18 to 65 years of age.
* HIV-1 infected.
* On a stable antiretroviral regimen for greater than or equal to 3 months.
* Available for clinical follow-up through the last study visit.
* Based on history and examination, must be in general good health with no evidence of clinically significant lab abnormalities and without additional clinically significant medical conditions as per exclusion criteria.
* Willing to maintain or establish a relationship with a primary health care provider for medical management of HIV infection while participating in the study.
* Willing to have blood samples collected, stored indefinitely, and used for research purposes.
* Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
* Laboratory tests assessing individual's health will be conducted within 84 days prior to enrollment and values must meet the following criteria:

  1. White blood cell count (WBC) 2,500-12,000/mm^3;
  2. WBC differential either within institutional normal range or accompanied by approval of the Principal Investigator (PI) or designee;
  3. Platelets = 125,000-400,000/mm^3;
  4. Hemoglobin greater than or equal to 10.0 gm/dL;
  5. Creatinine less than or equal to 1.25 x upper limit of normal (ULN);
  6. Alanine aminotransferase (ALT) less than or equal to 1.1 x ULN;
  7. Aspartate aminotransferase (AST) less than or equal to 1.1 x ULN; and,
  8. Viral Load (VL) less than or equal to 50 copies/mL and a CD4 count greater than or equal to 300/mcL (microliter).

     Male-Specific Criteria:
* Males must agree to use condoms for all sexual activity of any reproductive potential for 52 weeks after receiving the study product.

Female-Specific Criteria:

* If a woman is sexually active with a male partner and has no history of hysterectomy, tubal ligation or menopause, she must agree to use either a prescription birth control method or a barrier birth control method from the time of study enrollment through study Week 52, or to be monogamous with a partner who has had a vasectomy.
* Negative beta-HCG (human chorionic gonadotropin) pregnancy test (urine or serum) on day of enrollment for women presumed to be of reproductive potential.

EXCLUSION CRITERIA:

A volunteer would have been excluded if one or more of the following conditions applied:

* Previous receipt of monoclonal antibody whether licensed or investigational.
* Previous receipt of gene therapy product.
* Ongoing AIDS-related opportunistic infection (including oral thrush).
* Active injection drug use or active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* A titer of pre-existing antibodies to AAV8 capsid is greater than 1:90.
* Weight > 115 kg for Group 3 participants only.
* History of a severe allergic reaction with generalized urticaria, angioedema or anaphylaxis within the 2 years prior to enrollment that has a reasonable risk of recurrence.
* Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
* Active liver disease such as chronic hepatitis.
* Hypertension that is not well controlled by medication.
* Woman who is breast-feeding or planning to become pregnant during the study participation.
* Receipt of any investigational study agent within 28 days prior to enrollment.
* Current infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
* Any other chronic or clinically significant medical condition that in the opinion of investigator would jeopardize the safety or rights of the volunteer, including, but not limited to: diabetes mellitus type I; OR clinically significant forms of asthma, autoimmune disease, psychiatric disorders, heart disease, or cancer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2026-08-08 (Estimated); Study Completion 2026-08-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Casazza, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) is not shared because it has limited value in a small phase 1 trial. We instead report non-IPD data as required in ClinicalTrials.gov.

REFERENCES:
- [Background] Lynch RM, Boritz E, Coates EE, DeZure A, Madden P, Costner P, Enama ME, Plummer S, Holman L, Hendel CS, Gordon I, Casazza J, Conan-Cibotti M, Migueles SA, Tressler R, Bailer RT, McDermott A, Narpala S, O'Dell S, Wolf G, Lifson JD, Freemire BA, Gorelick RJ, Pandey JP, Mohan S, Chomont N, Fromentin R, Chun TW, Fauci AS, Schwartz RM, Koup RA, Douek DC, Hu Z, Capparelli E, Graham BS, Mascola JR, Ledgerwood JE; VRC 601 Study Team. Virologic effects of broadly neutralizing antibody VRC01 administration during chronic HIV-1 infection. Sci Transl Med. 2015 Dec 23;7(319):319ra206. doi: 10.1126/scitranslmed.aad5752. PMID 26702094
- [Background] Balazs AB, Ouyang Y, Hong CM, Chen J, Nguyen SM, Rao DS, An DS, Baltimore D. Vectored immunoprophylaxis protects humanized mice from mucosal HIV transmission. Nat Med. 2014 Mar;20(3):296-300. doi: 10.1038/nm.3471. Epub 2014 Feb 9. PMID 24509526
- [Result] Casazza JP, Cale EM, Narpala S, Yamshchikov GV, Coates EE, Hendel CS, Novik L, Holman LA, Widge AT, Apte P, Gordon I, Gaudinski MR, Conan-Cibotti M, Lin BC, Nason MC, Trofymenko O, Telscher S, Plummer SH, Wycuff D, Adams WC, Pandey JP, McDermott A, Roederer M, Sukienik AN, O'Dell S, Gall JG, Flach B, Terry TL, Choe M, Shi W, Chen X, Kaltovich F, Saunders KO, Stein JA, Doria-Rose NA, Schwartz RM, Balazs AB, Baltimore D, Nabel GJ, Koup RA, Graham BS, Ledgerwood JE, Mascola JR; VRC 603 Study Team. Safety and tolerability of AAV8 delivery of a broadly neutralizing antibody in adults living with HIV: a phase 1, dose-escalation trial. Nat Med. 2022 May;28(5):1022-1030. doi: 10.1038/s41591-022-01762-x. Epub 2022 Apr 11. PMID 35411076
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-I-0030.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteers were recruited for the study at the NIH Clinical Center in Bethesda, Maryland, USA. Adults who were HIV infected but in general good health and had been taking the same HIV medicine for at least 3 months were enrolled.
Period: One Year Follow Up
Arm/Group | Group 1: AAV8-VRC07 (5 x 10^10 vg/kg IM) | Group 2: AAV8-VRC07 (5 x 10^11 vg/kg IM) | Group 3: AAV8-VRC07 (2.5 x 10^12 vg/kg IM)
Started | 3 | 3 | 4
Received Study Product | 3 | 3 | 4
Completed (Participants who completed one year of study visits.) | 3 | 3 | 4
Not Completed | 0 | 0 | 0
Period: Five Year Long Term Follow Up
Arm/Group | Group 1: AAV8-VRC07 (5 x 10^10 vg/kg IM) | Group 2: AAV8-VRC07 (5 x 10^11 vg/kg IM) | Group 3: AAV8-VRC07 (2.5 x 10^12 vg/kg IM)
Started | 3 | 3 | 4
Completed (Participants who completed 5 years of the study per protocol as of May 2023) | 2 | 0 | 0
Not Completed | 1 | 3 | 4
Not completed — Long Term Follow Up Ongoing | 1 | 2 | 4
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Population included all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: AAV8-VRC07 (5 x 10^10 vg/kg IM) | Group 2: AAV8-VRC07 (5 x 10^11 vg/kg IM) | Group 3: AAV8-VRC07 (2.5 x 10^12 vg/kg IM) | Total
Number analyzed (Participants) | 3 | 3 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] — Age represents age at enrollment day.
  years | 50.7 (12.9) | 34.7 (15.5) | 43.0 (12.8) | 42.8 (13.7)
Age, Customized [Count of Participants; unit: Participants] — Age represents age at enrollment day.
  Participants
    21-30 years | 0 | 2 | 0 | 2
    31-40 years | 1 | 0 | 2 | 3
    41-50 years | 0 | 0 | 0 | 0
    51-60 years | 2 | 1 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 2
  Male | 3 | 3 | 2 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 1 | 3 | 5
  White | 2 | 2 | 1 | 5
  Hispanic/Latino | 0 | 0 | 1 | 1
  Non-Hispanic/Latino | 3 | 3 | 3 | 9
Weight (kg) [Mean (Standard Deviation); unit: kg] — Weight represents weight from enrollment evaluation.
  kg | 75.5 (8.6) | 74.5 (1.6) | 83.1 (8.8) | 78.2 (7.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms Within 7 Days of AAV8-VRC07 Product Administration
Description: Participants recorded the occurrence of solicited symptoms on a diary card for 7 days after study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Local Symptom" is the number of participants reporting any local symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases, Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1.
Time Frame: 7 days after AAV8-VRC07 product administration, at approximately Week 1
Population: Population included all enrolled participants who received AAV8-VRC07 and provided safety data (via diary card).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: AAV8-VRC07 (5 x 10^10 vg/kg IM) | Group 2: AAV8-VRC07 (5 x 10^11 vg/kg IM) | Group 3: AAV8-VRC07 (2.5 x 10^12 vg/kg IM)
Number analyzed (Participants) | 3 | 3 | 4
Participants
  Pain/Tenderness: None | 3 | 3 | 0
  Pain/Tenderness: Mild | 0 | 0 | 4
  Pain/Tenderness: Moderate | 0 | 0 | 0
  Pain/Tenderness: Severe | 0 | 0 | 0
  Swelling: None | 3 | 3 | 4
  Swelling: Mild | 0 | 0 | 0
  Swelling: Moderate | 0 | 0 | 0
  Swelling: Severe | 0 | 0 | 0
  Redness: None | 3 | 3 | 4
  Redness: Mild | 0 | 0 | 0
  Redness: Moderate | 0 | 0 | 0
  Redness: Severe | 0 | 0 | 0
  Any Local Symptom: None | 3 | 3 | 0
  Any Local Symptom: Mild | 0 | 0 | 4
  Any Local Symptom: Moderate | 0 | 0 | 0
  Any Local Symptom: Severe | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms Within 7 Days of AAV8-VRC07 Product Administration
Description: Participants recorded the occurrence of solicited symptoms on a diary card for 7 days after study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Systemic Symptom" is the number of participants reporting any systemic symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases, Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1.
Time Frame: 7 days after AAV8-VRC07 product administration, at approximately Week 1
Population: Population included all enrolled participants who received AAV8-VRC07 and provided safety data (via diary card).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: AAV8-VRC07 (5 x 10^10 vg/kg IM) | Group 2: AAV8-VRC07 (5 x 10^11 vg/kg IM) | Group 3: AAV8-VRC07 (2.5 x 10^12 vg/kg IM)
Number analyzed (Participants) | 3 | 3 | 4
Participants
  Malaise: None | 3 | 3 | 4
  Malaise: Mild | 0 | 0 | 0
  Malaise: Moderate | 0 | 0 | 0
  Malaise: Severe | 0 | 0 | 0
  Myalgia: None | 3 | 2 | 3
  Myalgia: Mild | 0 | 1 | 1
  Myalgia: Moderate | 0 | 0 | 0
  Myalgia: Severe | 0 | 0 | 0
  Headache: None | 3 | 3 | 2
  Headache: Mild | 0 | 0 | 2
  Headache: Moderate | 0 | 0 | 0
  Headache: Severe | 0 | 0 | 0
  Chills: None | 3 | 3 | 4
  Chills: Mild | 0 | 0 | 0
  Chills: Moderate | 0 | 0 | 0
  Chills: Severe | 0 | 0 | 0
  Nausea: None | 3 | 3 | 4
  Nausea: Mild | 0 | 0 | 0
  Nausea: Moderate | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0
  Temperature (Fever): None | 3 | 3 | 4
  Temperature (Fever): Mild | 0 | 0 | 0
  Temperature (Fever): Moderate | 0 | 0 | 0
  Temperature (Fever): Severe | 0 | 0 | 0
  Joint Pain: None | 3 | 3 | 4
  Joint Pain: Mild | 0 | 0 | 0
  Joint Pain: Moderate | 0 | 0 | 0
  Joint Pain: Severe | 0 | 0 | 0
  Any Systemic Symptom: None | 3 | 2 | 2
  Any Systemic Symptom: Mild | 0 | 1 | 2
  Any Systemic Symptom: Moderate | 0 | 0 | 0
  Any Systemic Symptom: Severe | 0 | 0 | 0

3. Primary Outcome: Number of Participants With One or More Unsolicited Non-Serious Adverse Events (AEs) Following AAV8-VRC07 Product Administration
Description: Unsolicited adverse event (AE) data collection included AEs of all severities from the date of product administration through the Day 56 (8 weeks) post-product administration visit. After the Day 56 (8 weeks) post-product administration visit, only serious AEs (SAEs reported as a separate outcome and in the AE module) and new chronic medical conditions that require ongoing medical management (reported as a separate outcome) will be recorded through the last study visit. The relationship between a non-serious AE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 through 8 weeks after AAV8-VRC07 product administration
Population: Population included all enrolled participants who received AAV8-VRC07 and had safety data collected (via clinical assessment and/or lab results).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: AAV8-VRC07 (5 x 10^10 vg/kg IM) | Group 2: AAV8-VRC07 (5 x 10^11 vg/kg IM) | Group 3: AAV8-VRC07 (2.5 x 10^12 vg/kg IM)
Number analyzed (Participants) | 3 | 3 | 4
Participants
  Related to Study Product | 1 | 0 | 1
  Unrelated to Study Product | 1 | 2 | 1
  Total Number of Participants who had One or More Non-Serious Unsolicited AE after AAV8-VRC07 Given | 2 | 2 | 2

4. Primary Outcome: Number of Participants With Abnormal Laboratory Measures of Safety Following AAV8-VRC07 Product Administration
Description: Abnormal laboratory results recorded as unsolicited adverse events (AEs) are summarized. Safety lab parameters included hematology (hemoglobin, hematocrit, mean corpuscular volume (MCV), platelets, and neutrophil, lymphocyte, monocyte, eosinophil and basophil counts) and chemistry (alanine aminotransferase (ALT), aspartate aminotransferase (AST) and creatinine). Complete Blood Count (CBC) with differential and chemistry (ALT, AST and creatinine) results were collected at different timepoints throughout the study per the protocol's schedule of evaluations. Institutional laboratory normal ranges as well as the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1 were used.
Time Frame: Day 0 through 8 weeks after AAV8-VRC07 product administration
Population: Population includes all enrolled participants who received AAV8-VRC07 and have or will have safety data collected via laboratory results.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: AAV8-VRC07 (5 x 10^10 vg/kg IM) | Group 2: AAV8-VRC07 (5 x 10^11 vg/kg IM) | Group 3: AAV8-VRC07 (2.5 x 10^12 vg/kg IM)
Number analyzed (Participants) | 3 | 3 | 4
Participants
  Aspartate aminotransferase (AST) | 2 | 0 | 0
  Creatinine | 1 | 0 | 2
  Number of Participants with one or more Abnormal Laboratory Results AE Related to Study Product | 1 | 0 | 1
  Number of Participants with one or more Abnormal Laboratory Results AE Unrelated to Study Product | 1 | 0 | 1
  Total Number of Participants who had Any Abnormal Laboratory Results Reported as AEs | 2 | 0 | 2

5. Primary Outcome: Geometric Mean Endpoint Titer of Anti-AAV8 Antibodies
Description: Anti-AAV8 antibodies were analyzed by enzyme-linked immunosorbent assay (ELISA) using a vector-matched AAV8 capsid as the capture agent. Group geometric means and 95% confidence intervals (CIs) for the endpoint titers for the AAV8 ELISA assay are reported at baseline, week 12 for the peak response, and week 44 for durability. Values below the lower limit of detection (LOD) were imputed to the lower LOD (30) and values above the assay upper LOD were imputed to the upper LOD (21870).
Time Frame: Day 0 through 44 Weeks after AAV8-VRC07 product administration
Population: Population included all enrolled participants who received AAV8-VRC07.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1: AAV8-VRC07 (5 x 10^10 vg/kg IM) | Group 2: AAV8-VRC07 (5 x 10^11 vg/kg IM) | Group 3: AAV8-VRC07 (2.5 x 10^12 vg/kg IM)
Number analyzed (Participants) | 3 | 3 | 4
titer
  Baseline, Week 0 (Visit 02) | 30 [NA to NA] — Values below the lower limit of detection (LOD) were imputed to the lower LOD (30) with no 95% CI indicated as (NA). | 30 [NA to NA] — Values below the lower limit of detection (LOD) were imputed to the lower LOD (30) with no 95% CI indicated as (NA). | 156 [84 to 290]
  Week 12 (Visit 14) | 5055 [2466 to 10361] | 10514 [5129 to 21552] | 21870 [21870 to 21870]
  Week 44 (Visit 25) | 5055 [1203 to 21238] | 7290 [2103 to 25272] | 21870 [21870 to 21870]

6. Primary Outcome: Number of Participants Who Attained A 50 mcg/mL VRC07 Serum Concentration
Description: In order to determine the optimal AAV8-VRC07 dose, participants must have attained a 50 mcg/mL VRC07 Serum Concentration. If no participants attained at least 50 mcg/mL VRC07 serum concentration, then the optimal AAV8-VRC07 dose cannot be determined.
Time Frame: Day 0 through 52 Weeks after AAV8-VRC07 product administration
Population: Population included all enrolled participants who received AAV8-VRC07.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: AAV8-VRC07 (5 x 10^10 vg/kg IM) | Group 2: AAV8-VRC07 (5 x 10^11 vg/kg IM) | Group 3: AAV8-VRC07 (2.5 x 10^12 vg/kg IM)
Number analyzed (Participants) | 3 | 3 | 4
Participants | 0 | 0 | 0

7. Primary Outcome: Geometric Mean Concentration of VRC07 Serum Antibodies (PK ELISA)
Description: For the pharmacokinetic (PK) primary outcome analysis, PK ELISA detected VRC07 serum antibodies in mcg/mL, using the VRC01 anti-idiotype Fab specific 5C9 monoclonal antibody (mAb). Only visits that had detectable PK ELISA concentrations for any participant are reported. Results are reported in group geometric mean mcg/mL concentrations with 95% CIs. The protocol specifies that a more sensitive assay can also be used; the more sensitive Singulex assay results are reported later in the secondary outcome measure. Values below the lower limit of detection (LOD) were imputed to the lower LOD (1 mcg/mL) with no 95% CI.
Time Frame: Day 0 through 52 Weeks after AAV8-VRC07 product administration
Population: Population included all enrolled participants who received AAV8-VRC07.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | Group 1: AAV8-VRC07 (5 x 10^10 vg/kg IM) | Group 2: AAV8-VRC07 (5 x 10^11 vg/kg IM) | Group 3: AAV8-VRC07 (2.5 x 10^12 vg/kg IM)
Number analyzed (Participants) | 3 | 3 | 4
mcg/mL
  Week 28 (Visit 21) | 1 [NA to NA] — Values below the lower limit of detection (LOD) were imputed to the lower LOD (1 mcg/mL) with no 95% CI indicated as (NA). | 1.10 [0.89 to 1.34] | 1 [NA to NA] — Values below the lower limit of detection (LOD) were imputed to the lower LOD (1 mcg/mL) with no 95% CI indicated as (NA).
  Week 36 (Visit 23) | 1 [NA to NA] — Values below the lower limit of detection (LOD) were imputed to the lower LOD (1 mcg/mL) with no 95% CI indicated as (NA). | 1.08 [0.92 to 1.25] | 1 [NA to NA] — Values below the lower limit of detection (LOD) were imputed to the lower LOD (1 mcg/mL) with no 95% CI indicated as (NA).
  Week 44 (Visit 25) | 1 [NA to NA] — Values below the lower limit of detection (LOD) were imputed to the lower LOD (1 mcg/mL) with no 95% CI indicated as (NA). | 1.04 [0.96 to 1.12] | 1 [NA to NA] — Values below the lower limit of detection (LOD) were imputed to the lower LOD (1 mcg/mL) with no 95% CI indicated as (NA).
  Week 52 (Visit 27) | 1 [NA to NA] — Values below the lower limit of detection (LOD) were imputed to the lower LOD (1 mcg/mL) with no 95% CI indicated as (NA). | 1.42 [0.41 to 2.82] | 1 [NA to NA] — Values below the lower limit of detection (LOD) were imputed to the lower LOD (1 mcg/mL) with no 95% CI indicated as (NA).

8. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) Following AAV8-VRC07 Product Administration
Description: SAEs are recorded from receipt of study product through the last expected study visit at Year 5 (260 weeks). The relationship between a SAE and the study product is assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 through 5 Years (260 weeks) after AAV8-VRC07 product administration
Reporting Status: Not Posted, anticipated posting 2026-08

9. Primary Outcome: Number of Participants With New Chronic Medical Conditions Following AAV8-VRC07 Product Administration
Description: New chronic medical conditions are recorded from receipt of study product through the last expected study visit at Year 5 (260 weeks). The relationship between a new chronic medical condition and the study product is assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 through 5 Years (260 weeks) after AAV8-VRC07 product administration
Reporting Status: Not Posted, anticipated posting 2026-08

10. Primary Outcome: Number of Participants Who Produced VRC07 Anti-drug Antibodies (ADA)
Description: A three-tiered assay was used for ADA evaluation. The tier 1 screening assay measures specific and non-specific binding of serum proteins to VRC07 and the assay membrane. The tier 2 assay is a qualitative competition assay in which exogenously added VRC07 removes any VRC07-binding proteins from the serum prior to the binding assay. If the addition of the exogenous VRC07 results in a reduction of signal, the specificity of VRC07 binding is confirmed. The tier 3 assay is a qualitative assay that assesses the ability of VRC07-binding serum protein to prevent VRC07-mediated neutralization of an HIV pseudovirus in vitro. Only samples positive for a tier will be analyzed in subsequent tiers.
Time Frame: Day 0 through 5 Years (260 weeks) after AAV8-VRC07 product administration
Reporting Status: Not Posted, anticipated posting 2026-08

11. Secondary Outcome: Geometric Mean Value of CD4 Cell Counts
Description: The clinical effects of pAAV8-VRC07 on cluster of differentiation 4 (CD4) cell count were assessed. CD4 Cell Count (cells/mL) shown as reported by the Clinical Center serology lab. Values are reported as group geometric means and 95% CIs.
Time Frame: Day 0 through 44 Weeks after AAV8-VRC07 product administration
Population: Population included all enrolled participants who received AAV8-VRC07.
Measure: Geometric Mean (95% Confidence Interval); unit: cells/mL
Arm/Group | Group 1: AAV8-VRC07 (5 x 10^10 vg/kg IM) | Group 2: AAV8-VRC07 (5 x 10^11 vg/kg IM) | Group 3: AAV8-VRC07 (2.5 x 10^12 vg/kg IM)
Number analyzed (Participants) | 3 | 3 | 4
cells/mL
  Baseline, Week 0 (Visit 02) | 499 [447 to 557] | 599 [339 to 1057] | 551 [404 to 750]
  Week 12 (Visit 14) | 519 [446 to 604] | 595 [389 to 908] | 557 [463 to 669]
  Week 25 (Visit 44) | 574 [402 to 820] | 629 [547 to 723] | 548 [412 to 729]

12. Secondary Outcome: Viral Load
Description: The clinical effects of pAAV8-VRC07 on viral load were assessed. Viral Load is expressed in polymerase chain reaction (PCR) copies/mL, as reported by the Clinical Center serology lab. Values below the limit of quantification (<20 copies/mL) or none detected were imputed to 10 copies/mL. Results are displayed as median(range).
Time Frame: Day 0 through 44 Weeks after AAV8-VRC07 product administration
Population: Population included all enrolled participants who received AAV8-VRC07.
Measure: Median (Full Range); unit: copies/mL
Arm/Group | Group 1: AAV8-VRC07 (5 x 10^10 vg/kg IM) | Group 2: AAV8-VRC07 (5 x 10^11 vg/kg IM) | Group 3: AAV8-VRC07 (2.5 x 10^12 vg/kg IM)
Number analyzed (Participants) | 3 | 3 | 4
copies/mL
  Baseline, Week 0 (Visit 02) | 10 [NA to 23] — Values below the lower limit of detection (LOD, 20 copies/mL) were imputed as 10 copies/mL with no range indicated as (NA). | 10 [NA to NA] — Values below the lower limit of detection (LOD, 20 copies/mL) were imputed as 10 copies/mL with no range indicated as (NA). | 10 [NA to NA] — Values below the lower limit of detection (LOD, 20 copies/mL) were imputed as 10 copies/mL with no range indicated as (NA).
  Week 12 (Visit 14) | 10 [NA to NA] — Values below the lower limit of detection (LOD, 20 copies/mL) were imputed as 10 copies/mL with no range indicated as (NA). | 10 [NA to NA] — Values below the lower limit of detection (LOD, 20 copies/mL) were imputed as 10 copies/mL with no range indicated as (NA). | 10 [NA to NA] — Values below the lower limit of detection (LOD, 20 copies/mL) were imputed as 10 copies/mL with no range indicated as (NA).
  Week 44 (Visit 25) | 10 [NA to NA] — Values below the lower limit of detection (LOD, 20 copies/mL) were imputed as 10 copies/mL with no range indicated as (NA). | 10 [NA to 30] — Values below the lower limit of detection (LOD, 20 copies/mL) were imputed as 10 copies/mL with no range indicated as (NA). | 10 [NA to 29] — Values below the lower limit of detection (LOD, 20 copies/mL) were imputed as 10 copies/mL with no range indicated as (NA).

13. Secondary Outcome: Concentration of VRC07 Serum Antibodies (Singulex Assay)
Description: The serum concentration of VRC07 at specified time intervals for 1 year after injection was determined, and if persistent, then every 6 months as long as there is detectable antibody in serum. The PK Singulex assay utilizes a microparticle-based immunoassay coupled with a fluorescent detection system to detect serum antibodies in the ng/mL range. Values below the limit of detection or none detected were set to 0.10 ng/mL; therefore, a value of 0.10 ng/mL means that the VRC07 concentration for that assay was below the limit of detection. Results are displayed as median(range).
Time Frame: Day 0 through 52 weeks after AAV8-VRC07 product administration
Population: Population includes all enrolled participants who received AAV8-VRC07.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Group 1: AAV8-VRC07 (5 x 10^10 vg/kg IM) | Group 2: AAV8-VRC07 (5 x 10^11 vg/kg IM) | Group 3: AAV8-VRC07 (2.5 x 10^12 vg/kg IM)
Number analyzed (Participants) | 3 | 3 | 4
ng/mL
  Baseline, Week 0 (Visit 02) | 0.10 [0.10 to 20.26] | 0.10 [0.10 to 1.06] | 9.69 [0.10 to 13.62]
  Week 6 (Visit 08) | 281.29 [71.06 to 401.70] | 216.71 [36.20 to 598.53] | 304.93 [37.04 to 1221.45]
  Week 24 (Visit 20): number analyzed (Participants) | 3 | 3 | 2
  Week 24 (Visit 20) | 374.63 [48.62 to 375.06] | 34.30 [5.85 to 413.50] | 908.01 [550.89 to 1265.14]
  Week 52 (Visit 27) | 316.29 [127.49 to 350.34] | 9.24 [0.10 to 711.83] | 354.26 [39.39 to 2469.31]

ADVERSE EVENTS:
Time Frame: Unsolicited adverse event (AE) data collection included AEs of all severities from the date of product administration through the Day 56 (8 weeks) visit. After the Day 56 visit, only serious AEs (SAEs) and new chronic medical conditions (NCMCs) that require ongoing medical management will be recorded through the last expected LTFU visit at Year 5 (260 weeks). After all data are collected, the data reported now for the Day 56 Time Frame will be updated to reflect all post-Day 56 SAEs and NCMCs.
Description: Solicited AEs collected through systematic assessment and unsolicited AEs collected through non-systematic assessment represent the number and percentage of participants reporting the event. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Arm/Group | Group 1: AAV8-VRC07 (5 x 10^10 vg/kg IM) | Group 2: AAV8-VRC07 (5 x 10^11 vg/kg IM) | Group 3: AAV8-VRC07 (2.5 x 10^12 vg/kg IM)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: AAV8-VRC07 (5 x 10^10 vg/kg IM) (N=3) | Group 2: AAV8-VRC07 (5 x 10^11 vg/kg IM) (N=3) | Group 3: AAV8-VRC07 (2.5 x 10^12 vg/kg IM) (N=4)
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Administration site pain (General disorders) | 0 | 0 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
The active phase of the study was completed on August 2, 2022 and data collection is complete for the majority of the outcome measures; therefore, those completed measures are being reported after one year of follow up. The primary outcomes for SAEs, NCMCs and VRC07 ADAs will be reported once all participants have completed the Year 5 LTFU study visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-02-18): https://cdn.clinicaltrials.gov/large-docs/02/NCT03374202/Prot_SAP_ICF_001.pdf